CLINICAL TRIAL: NCT01006408
Title: Pilot, Single Center, Randomized, Double Blind, Placebo Controlled, Single Crossover Treatment Trial Using Low Level Laser Therapy (LLLT) for Treatment of Chemotherapy Induced Peripheral Neuropathy
Brief Title: Treatment Trial Using Low Level Laser Therapy (LLLT) for Treatment of Chemotherapy Induced Peripheral Neuropathy
Acronym: LLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Nathalie Johnson, Principal investigator, Legacy Health System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LLLT-001
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Peripheral Neuropathy
Keywords: Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Level Laser (Active Comparator): Low Level Laser twice a week for 8 weeks
  Interventions: Procedure: Low Level Laser
- Placebo and Low Level Laser (Sham Comparator): Placebo twice a week for 4 weeks then crossover to Low Level Laser twice a week for 4 weeks
  Interventions: Procedure: Placebo followed by Low Level Laser

INTERVENTIONS:
Procedure: Low Level Laser — Low Level Laser twice a week for 8 weeks
  Arms: Low Level Laser
Procedure: Placebo followed by Low Level Laser — Placebo twice a week for 4 weeks then crossover to Low Level Laser twice a week for 4 weeks
  Arms: Placebo and Low Level Laser

SUMMARY:
The purpose of this research study is to determine if treatment with Low Level Laser Therapy (LLLT) is effective in treating the pain, numbness or tingling patients are experiencing following their chemotherapy. The investigators would also like to know the number of treatments that were needed in order to reduce their symptoms.

DETAILED DESCRIPTION:
LLLT is a technique of applying a low energy or low-level laser to tissue. It is used to trigger tissue to increase cellular production by giving off a low-level, or cold light energy. This low level energy passes through the skin, into the cell membrane producing a process called photobiostimulation. LLLT works by capturing and increasing the beneficial wavelengths of light. These lasers do not cut or burn, but instead penetrate into the skin. This process has multiple effects on cells and can enhance the body's natural regenerative functions. It can also stimulate the release of endorphins and collagen. Endorphins work as "natural pain relievers" and are produced by the body during strenuous workouts, excitement and pain. Collagen is a natural substance within body tissues.

This is a single center trial conducted at Legacy Health System. Twenty patients from Legacy Health System with chemo-induced peripheral neuropathy will be enrolled in this study. Arm 1 will receive LLLT twice a week for a total of eight weeks. Arm 2 will follow a crossover study design where patients will receive sham (fake) LLLT twice a week for the first four weeks, followed by true LLLT twice a week for four weeks, (total of 8 weeks). Each patient in Arm 2 will serve as his or her own comparison for the purpose of examining the effects of LLLT. Both arms will have a follow-up visit following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion > 18 years of age
2. Male or Female
3. History of Cancer
4. Naive to LLLT
5. Completed chemotherapy between > 2 weeks & < 12 weeks OR > 9 months OR (pain or tingling in the upper or lower extremities beginning in association with cancer chemotherapy agent and persisting for at lease 28 days following conclusion of the chemotherapy. Pain can be assessed 28 days or more after the conclusion of chemotherapy)
6. Not pregnant
7. Consents to study participation
8. English Speaking
9. Minimal ambulatory with walker/cane or independent for 50 feet
10. Symptoms of neuropathy, including paresthesias, numbness and/or tingling of feet, toes and/or hands, fingers

Exclusion Criteria:

1. < 18 years of age
2. Previous treatment with LLLT
3. Neuropathy before chemotherapy
4. Current use of any topical treatment, nerve blocks, implantable therapy, or peripheral nerve or spinal cord stimulation, and neurosurgical procedure for painful CIPN
5. Subject who will not agree to maintain systemic pain treatments at stable dosages during the conduct of the study.
6. Adjunctive analgesic therapy such as acupuncture, biofeedback, or herbal preparations that has not been stable for at least 2 weeks
7. Subjects receiving an unapproved experimental drug or biological agent within 30 days of the screening visit
8. Subjects unable to complete assessment forms
9. Wheelchair dependent or non-ambulatory
10. Clinically significant depression or dementia that, in the opinion of the investigator, may interfere with a subjects' adherence to the study protocol and/or the accurate and consistent reporting of pain.
11. ETOH abuse as determined by the investigator
12. Open skin lesions in the area where the LLLT will be applied
13. Pregnant or lactating
14. Refuse to consent to trial participation
15. < 2 or > 12 weeks post chemotherapy OR between > 12 weeks and < 9 months post chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Legacy Good Samaritan Medical Center, Portland, Oregon, United States